CLINICAL TRIAL: NCT03901469
Title: A Phase 2b Study of ZEN003694 in Combination With Talazoparib in Patients With Triple-Negative Breast Cancer
Brief Title: A Study of ZEN003694 and Talazoparib in Patients With Triple Negative Breast Cancer
Acronym: TNBC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Parts 1 and 2 and Expansion Cohort C were completed. Expansion Cohorts A and B were discontinued based on results from an interim futility analysis and not due to safety concerns.
Sponsor: Zenith Epigenetics (Industry)
Collaborators: Pfizer (Industry); Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZEN003694-004; 2018-003906-26 (EudraCT Number)
Record Dates: First submitted 2019-03-22; First posted 2019-04-03 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer
Keywords: TNBC; ZEN003694; ZEN-3694; Talazoparib; Breast Cancer; PARPi; poly ADP ribose polymerase; bromodomain; BETi
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 and Part 2 (Experimental): ZEN003694 will be administered PO QD with Talazoparib PO QD in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
  Interventions: Drug: ZEN003694; Drug: Talazoparib
- Expansion Cohort A - Combination Treatment in post-TROP2-ADC patients (Experimental): ZEN003694 will be administered PO QD with Talazoparib PO QD at the RP2D in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
  Interventions: Drug: ZEN003694; Drug: Talazoparib
- Expansion Cohort B - ZEN003694 Monotherapy (Experimental): ZEN003694 will be administered PO QD as monotherapy at the RP2D in 28-day cycles with the option to cross-over to combination treatment of ZEN003694 PO QD with Talazoparib PO QD at the time of disease progression (but no sooner than after 6 weeks of monotherapy). Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
  Interventions: Drug: ZEN003694
- Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve patients (Experimental): ZEN003694 will be administered PO QD with Talazoparib PO QD at the RP2D in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in China only.
  Interventions: Drug: ZEN003694; Drug: Talazoparib

INTERVENTIONS:
Drug: ZEN003694 — PO QD
  Other Names: ZEN-3694
Drug: Talazoparib — PO QD
  Other Names: Talzenna
  Arms: Expansion Cohort A - Combination Treatment in post-TROP2-ADC patients; Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve patients; Part 1 and Part 2

SUMMARY:
This is a two-part open label, non-randomized, Phase 2, study of ZEN003694 in combination with Talazoparib in patients with TNBC without germline mutations of BRCA1 or BRCA2. Part 1 is a dose escalation and Part 2 is a Simon 2-Stage design. There are 3 expansion cohorts: Expansion Cohort A (combination treatment in post-TROP2-ADC patients), Expansion Cohort B (ZEN003694 monotherapy), and Expansion Cohort C (combination treatment in TROP2-ADC-naive patients).

ELIGIBILITY:
Inclusion Criteria:

1. Females or males age ≥ 18 years (at time of signing informed consent)
2. Parts 1 and 2 only: Histologically confirmed metastatic or recurrent or locally advanced triple-negative breast cancer (estrogen receptor (ER) ≤10%; progesterone receptor (PR) ≤10%; and HER2 negative by immunohistochemistry (IHC) or fluorescent in situ hybridization (FISH)

   Expansion only: Histologically confirmed metastatic or recurrent, or locally advanced triple-negative breast cancer as defined by the most recent American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines.
3. Patient is not a candidate for endocrine based therapy, based on Investigator judgement
4. Have a history of progressive disease despite prior therapy
5. Part 1: Have had at least 1 prior cytotoxic chemotherapy.

   Part 2: Have had no more than 2 prior chemotherapy-inclusive regimens for locally advanced or metastatic disease, unless approved by the Sponsor (no limit on prior targeted anticancer therapies such as mechanistic target or rapamycin (mTOR) or CDK4/6 inhibitors, immune-oncology agents, tyrosine kinase inhibitors, or monoclonal antibodies against CTL4 or VEGF.)

   Expansion Cohort A (combination treatment in post-TROP2-ADC patients): Have received TROP2-ADC therapy for unresectable locally advanced or metastatic disease.

   Expansion Cohort B (ZEN003694 monotherapy): Have had at least 1 prior systemic therapy for locally advanced or metastatic disease which may or may not have included a TROP2-ADC.

   Expansion Cohort C (combination treatment in TROP2-ADC-naive patients): Have had at least 1 prior systemic therapy for locally advanced or metastatic disease and who have not received prior TROP2-ADC therapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Part 2 and Expansion only: Measurable disease per RECIST version 1.1

Exclusion Criteria:

1. Documented germline mutations of BRCA1 or BRCA2
2. Parts 1 and 2 only: Evidence of disease progression during platinum treatment either in the neoadjuvant or in the metastatic setting. For patients receiving platinum in the neoadjuvant setting, at least 6 months must have elapsed between the last dose of platinum-based treatment and enrollment
3. Part 2 only: Patients with inflammatory breast cancer
4. Current or anticipated use of medications known to be strong inhibitors or inducers of CYP3A4 or substrates of CYP1A2 with narrow therapeutic windows. Strong inhibitors, inducers or substrates must be discontinued at least 7 days prior to the first administration of study drug.
5. Current or anticipated use within 7 days prior to the first administration of study drug, or during the study, of strong P-gp inhibitors.
6. Use of oral Factor Xa inhibitors (i.e., rivaroxaban, apixaban, betrixaban, edoxaban otamixaban, letaxaban, eribaxaban) and Factor IIa inhibitors (i.e., dabigatran). Low molecular weight heparin is allowed
7. Prior anticancer therapy (chemotherapy, radiation, hormone therapy, immunotherapy or investigational agent) within 3 weeks from the start of study drug (except for nitrosoureas and mitomycin C within 6 weeks from start of study drug)
8. Parts 1 and 2 only: Radiation to >25% of the bone marrow
9. Treatment with a bone-targeted radionuclide within 6 weeks of first dose of study drug
10. Have previously received an investigational BET inhibitor (including previous participation in studies with the Sponsor's drug, ZEN003694); except for patients in Expansion Cohort B who received ZEN003694 monotherapy and are eligible to cross-over to combination treatment
11. Prior treatment with a PARP inhibitor
12. QTcF interval > 470 msec
13. Insufficient recovery (i.e., has not recovered to at least Grade 1) from prior treatment-related toxicities except for alopecia, fatigue and Grade 2 neuropathy
14. Non-healing wound, ulcer or bone fracture (not including a pathological bone fracture caused by a pre-existing pathological bone lesion)
15. Parts 1 and 2 only: Brain metastases not adequately treated and clinically stable (at the discretion of the Investigator) for at least 3 months prior to the start of study treatment, unless a shorter interval is approved by the Sponsor's Medical Monitor

    Expansion only: Progressive, symptomatic, or untreated brain metastases. CNS metastases treated definitively with surgery and/or radiation must be radiographically stable based on imaging at least 3 months after definitive treatment. CNS metastases requiring steroid doses equivalent to prednisone doses >10 mg daily or an increase in steroid doses due to CNS disease prior to consent are not eligible
16. Expansion only: Disease initially diagnosed with expression of estrogen receptor (ER) or progesterone receptor (PR) as ≥5%
17. Expansion only: Patients treated with prior endocrine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (8):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Kansas Cancer Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Tennessee Oncology (Sarah Cannon), Nashville, Tennessee
  - MD Anderson, Houston, Texas
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - UZ Leuven, Leuven
- China (7):
  - The First Affiliated Hosptial of Bengbu Medical College, Bengbu, Anhui
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - Affliated Hospital of Jining Medical University, Jining, Shandong
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Tianjing Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
- Spain (2):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - START Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kharenko OA, Patel RG, Calosing C, van der Horst EH. Combination of ZEN-3694 with CDK4/6 inhibitors reverses acquired resistance to CDK4/6 inhibitors in ER-positive breast cancer. Cancer Gene Ther. 2022 Jun;29(6):859-869. doi: 10.1038/s41417-021-00375-9. Epub 2021 Aug 12. PMID 34385584

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at nineteen investigational sites in the United States (eight), Belgium (two), Spain (two), and China (seven) between June 2019 and March 2024
Pre-assignment Details: 115 participants were enrolled and treated in the study.
Groups:
- Part 1 Dose Escalation: Cohort 1: ZEN003694 48 mg PO QD with Talazoparib 1 mg PO QD in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
- Part 1 Dose Escalation: Cohort 2; Part 2 Stages 1 & 2: ZEN003694 48 mg PO QD with Talazoparib 0.75 mg PO QD in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
- Part 1 Dose Escalation: Cohort 3: ZEN003694 36 mg PO QD with Talazoparib 1 mg PO QD in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
- Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients: ZEN003694 48 mg PO QD with Talazoparib 0.75 mg PO QD (RP2D) in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
- Expansion Cohort B - ZEN003694 Monotherapy: ZEN003694 48 mg PO QD as monotherapy at the in 28-day cycles with the option to cross-over to combination treatment of ZEN003694 48 mg PO QD with 0.75 mg Talazoparib PO QD at the time of disease progression (but no sooner than after 6 weeks of monotherapy). Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
- Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients: ZEN003694 48 mg PO QD with Talazoparib PO QD (RP2D) in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in China only.
Period: Overall Study
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 2 Stages 1 & 2 | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients | Expansion Cohort B - ZEN003694 Monotherapy | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients
Started | 6 | 8 | 3 | 42 | 21 | 3 | 32
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 8 | 3 | 42 | 21 | 3 | 32
Not completed — Radiographic Progression | 4 | 6 | 3 | 30 | 7 | 2 | 11
Not completed — Clinical Progression | 0 | 2 | 0 | 7 | 6 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 9
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 8
Not completed — Death | 0 | 0 | 0 | 3 | 5 | 0 | 1
Not completed — Termination of study by sponsor | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated safety population consisted of all treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 2 Stages 1 & 2 | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients | Expansion Cohort B - ZEN003694 Monotherapy | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients | Total
Number analyzed (Participants) | 6 | 8 | 3 | 42 | 21 | 3 | 32 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (14.77) | 52.8 (11.72) | 59.3 (4.04) | 52.2 (12.09) | 49.2 (11.74) | 55.3 (10.12) | 54.9 (10.70) | 53.0 (11.57)
Age, Continuous [Median (Full Range); unit: years] | 55 [40 to 74] | 53 [31 to 69] | 57 [57 to 64] | 51.5 [28 to 80] | 49 [32 to 68] | 50 [49 to 67] | 55 [34 to 77] | 52 [28 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 3 | 42 | 21 | 3 | 32 | 115
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 6
  Not Hispanic or Latino | 5 | 7 | 2 | 40 | 18 | 3 | 20 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 12 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 3 | 0 | 31 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 5
  White | 5 | 6 | 3 | 38 | 14 | 2 | 0 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 3 | 2 | 1 | 1 | 8
Height [Mean (Standard Deviation); unit: cm] — Population: Data not available for all study participants
  cm
    number analyzed (Participants) | 6 | 8 | 3 | 40 | 18 | 3 | 32 | 110
    (all) | 164.60 (5.088) | 163.74 (5.882) | 165.00 (3.606) | 162.42 (6.730) | 163.66 (5.872) | 165.67 (16.512) | 157.2 (4.84) | 161.48 (6.07)
Height [Median (Full Range); unit: cm] — Population: Data not available for all study participants
  cm
    number analyzed (Participants) | 6 | 8 | 3 | 40 | 18 | 3 | 32 | 110
    (all) | 164.15 [158.0 to 170.0] | 166.35 [150.0 to 167.6] | 164.0 [162.0 to 169.0] | 164.5 [148.5 to 174.0] | 165.2 [150.2 to 170.2] | 175.2 [146.6 to 175.2] | 157.5 [146 to 166] | 162.5 [146 to 175.2]
Weight [Mean (Standard Deviation); unit: kg] | 76.32 (21.731) | 79.35 (23.396) | 74.00 (18.672) | 67.25 (12.804) | 72.98 (14.325) | 62.30 (5.726) | 61.55 (10.212) | 68.07 (13.531)
Weight [Median (Full Range); unit: kg] | 69.9 [55.7 to 116.0] | 72.9 [59.0 to 124.7] | 66.8 [60.0 to 95.2] | 66.0 [44.9 to 99.5] | 77.7 [47.3 to 93.0] | 64.5 [55.8 to 66.6] | 59.0 [41.5 to 80.0] | 65.4 [41.5 to 124.7]
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Data not available for all study participants
  kg/m^2
    number analyzed (Participants) | 6 | 8 | 3 | 40 | 18 | 3 | 32 | 110
    (all) | 28.50 (9.682) | 29.47 (7.961) | 27.01 (5.563) | 25.84 (4.710) | 27.01 (4.917) | 22.89 (2.683) | 24.928 (4.057) | 26.13 (5.029)
BMI [Median (Full Range); unit: kg/m^2] — Population: Data not available for all study participants
  kg/m^2
    number analyzed (Participants) | 6 | 8 | 3 | 40 | 18 | 3 | 32 | 110
    (all) | 24.61 [21.4 to 46.5] | 27.65 [21.1 to 45.4] | 24.84 [22.9 to 33.3] | 25.90 [19.1 to 40.1] | 27.16 [19.0 to 34.6] | 21.70 [21.0 to 26.0] | 25.195 [17.73 to 33.30] | 25.57 [17.73 to 46.5]
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work)
  2. - Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  4. - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  5. - Dead
  Participants
    ECOG 0 | 4 | 4 | 2 | 26 | 14 | 1 | 15 | 66
    ECOG 1 | 2 | 4 | 1 | 16 | 6 | 2 | 17 | 48
    ECOG 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1 and Part 2: Number of Participants With Treatment-related Adverse Events (AE) and Treatment-related Serious Adverse Events (SAE)
Time Frame: Cycle 1 Day 1 to 30 days post last dose (each cycle is 28 days) up to 22 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 2 Stages 1 & 2
Number analyzed (Participants) | 6 | 8 | 3 | 42
Participants
  Patients Reporting at least one TEAE related to study treatment | 6 | 8 | 3 | 41
  Patients reporting at least one Serious TEAE related to study treatment | 2 | 1 | 0 | 4

2. Primary Outcome: Part 1: Number of Participants With Dose-limiting Toxicities (DLT)
Description: Determination of DLT will be made during the first 28 days of treatment (i.e., Cycle 1) in the dose escalation phase. A DLT is defined as a clinically significant AE or laboratory abnormality that is considered possibly, probably or definitely related to study drug.
Time Frame: Cycle 1, Up to 1 month
Measure: Number; unit: participants
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3
Number analyzed (Participants) | 6 | 8 | 3
participants
  Platelet count decreased | 1 | 1 | 0
  Platelet count decreased/ Fatigue | 1 | 0 | 0

3. Primary Outcome: Part 2: Clinical Benefit Rate (CBR)
Description: Percentage of patients with a best overall response of confirmed complete response (CR), partial response (PR), or stable disease (SD ≥ 4 cycles) by RECIST v1.1
Time Frame: From screening up to 18 months
Population: Patients who have received at least 3 weeks of per-protocol treatment during Cycle 1, or <3 weeks of treatment in Cycle 1 because of a DLT, will comprise the Efficacy Population. Patients who were determined to be "unevaluable" during Cycle 1 by the Sponsor and Investigator will not be included in the Efficacy Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2 Stages 1 & 2
Number analyzed (Participants) | 37
Percentage of participants | 32.4

4. Primary Outcome: Expansion Cohort A: Objective Response Rate (ORR) by RECIST v1.1 (CR or PR)
Description: Percentage of participants with a confirmed complete response (CR) or partial response (PR) by RECIST 1.1
Time Frame: From screening up to 18 months
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients
Number analyzed (Participants) | 14
Percentage of participants | 0

5. Secondary Outcome: Part 1, Expansion Cohorts A and C: Clinical Benefit Rate (CBR)
Description: Percentage of participants with a confirmed complete response (CR), partial response (PR), or stable disease (SD ≥ 4 cycles) by RECIST 1.1
Time Frame: From screening up to 18 months
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Groups:
- Part 1 Dose Escalation - Cohort 1: ZEN003694 48 mg PO QD with Talazoparib 1 mg PO QD in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
Arm/Group | Part 1 Dose Escalation - Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients
Number analyzed (Participants) | 6 | 6 | 3 | 14 | 18
Percentage of participants | 33.3 | 66.7 | 33.3 | 0 | 11.1

6. Secondary Outcome: Part 1, Part 2, and Expansion Cohort C: Objective Response Rate (ORR)
Description: Percentage of participants with a confirmed complete response (CR) or partial response (PR) by RECIST 1.1
Time Frame: From screening up to 18 months
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 2 Stages 1 & 2 | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients
Number analyzed (Participants) | 6 | 6 | 3 | 37 | 18
Percentage of participants | 33.3 | 16.7 | 33.3 | 21.6 | 5.6

7. Secondary Outcome: Part 2, Expansion Cohorts A and C: Safety Profile of ZEN003694 in Combination With Talazoparib.
Description: Incidence of Treatment-related Adverse Events (AE) and Treatment-related Serious Adverse Events (SAE) in Part 2, Expansion Cohorts A and C
Time Frame: From screening up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Stages 1 & 2 | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients
Number analyzed (Participants) | 41 | 21 | 32
Participants
  Patients reporting at least one TEAE related to study treatment | 41 | 19 | 32
  Patients reporting at least one Serious TEAE related to study treatment | 4 | 1 | 13

8. Secondary Outcome: Part 1, Part 2, Expansion Cohorts A & C: Evaluate Median Progression-free Survival
Description: Median progression-free survival is the time from randomization to documented disease progression or death
Time Frame: From screening up to 18 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 Dose Escalation - Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 2 Stages 1 & 2 | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients
Number analyzed (Participants) | 6 | 6 | 3 | 37 | 14 | 18
months | 5.42 [NA to 9.2] — Insufficient sample size for software to calculate the lower confidence interval limit for median PFS | 5.06 [NA to NA] — Insufficient sample size for software to calculate the lower and upper confidence interval limit for median PFS | 1.51 [NA to 14.62] — Insufficient sample size for software to calculate the lower confidence interval limit for median PFS | 3.25 [1.84 to 5.09] | 1.38 [1.15 to 2.73] | 1.71 [1.41 to 3.88]

9. Secondary Outcome: Part 2, Expansion Cohorts A and C: Evaluate Duration of Response (DOR)
Description: For subjects with a confirmed response of PR or CR, duration of response is measured from the date of the first response until the time that overall disease progression (radiographic progressive disease or clinical deterioration) or death is documented.
Time Frame: From screening up to 18 months
Population: Participants with a confirmed response of PR or CR are included for the duration of response analysis
Measure: Median (Full Range); unit: months
Arm/Group | Part 2 Stages 1 & 2 | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients
Number analyzed (Participants) | 8 | 0 | 1
months | 4.7 [1.8 to 16.6] |  | 8.3

10. Secondary Outcome: Part 1 and Part 2: Measure the Pharmacokinetic Parameter (PK) of Cmax of ZEN003694 and ZEN003791 (Active Metabolite)
Description: Cmax is defined as the maximum or peak plasma concentration of drug (calculated from samples taken over a 4-hour or 8-hour time period). Cmax(0-8h) was calculated for Cycle 1, Day 1. Cmax(0-4h) was calculated for Cycle 2, Day 1. Pre-dose is time 0 for calculations.
Time Frame: Part 1: Cycle 1 Day 1: Pre-dose, 15 min, 30 min, 1 hour, 2 hour, 4 hour, 6 hour, and 8 hours post-dose. Parts 1 & 2: Cycle 2 Day 1: Pre-dose, 1 hour, 2 hour, and 4 hours post-dose. (cycles are 28 days)
Population: Part 1 (All evaluable participants): C1D1; Parts 1 & 2 (All evaluable participants): C2D1
Measure: Geometric Mean (Standard Error); unit: ng/ML
Groups:
- Part 2 - Stages 1 and 2: ZEN003694 48 mg PO QD with Talazoparib 0.75 mg PO QD in 28-day cycles. Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 2 - Stages 1 and 2
Number analyzed (Participants) | 6 | 8 | 3 | 28
ng/ML
  Cycle 1 Day 1 - ZEN003694: number analyzed (Participants) | 6 | 8 | 3 | 0
  Cycle 1 Day 1 - ZEN003694 | 406 (166) | 407 (104) | 143 (119) |
  Cycle 2 Day 1 - ZEN003694: number analyzed (Participants) | 4 | 2 | 3 | 28
  Cycle 2 Day 1 - ZEN003694 | 217 (154) | 465 (158) | 401 (174) | 513 (196)
  Cycle 1 Day 1 - ZEN003791: number analyzed (Participants) | 6 | 8 | 3 | 0
  Cycle 1 Day 1 - ZEN003791 | 202 (60) | 187 (65) | 66 (30) |
  Cycle 2 Day 1 - ZEN003791: number analyzed (Participants) | 4 | 2 | 3 | 28
  Cycle 2 Day 1 - ZEN003791 | 88 (30) | 242 (81) | 218 (80) | 285 (127)

11. Secondary Outcome: Part 1 and Part 2: Measure the Pharmacokinetic (PK) Parameter of Combined AUC(0-4h or 0-8h) of ZEN003694 and ZEN003791 (Active Metabolite)
Description: AUC(0-4h or 0-8h) is defined as the area under the curve (plasma concentration of drug calculated from samples taken over a 4-hour or 8-hour time period). AUC(0-8h) was calculated for Cycle 1, Day 1. AUC(0-4h) was calculated for Cycle 2, Day 1. Pre-dose is time 0 for calculations.
Time Frame: as for outcome 10
Population: Part 1 (All evaluable participants): C1D1; Parts 1 & 2 (All evaluable participants): C2D1
Measure: Geometric Mean (Standard Error); unit: ng*h/mL
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 2 - Stages 1 and 2
Number analyzed (Participants) | 6 | 8 | 3 | 28
ng*h/mL
  AUC(0-8h) Cycle 1 Day 1: number analyzed (Participants) | 6 | 8 | 3 | 0
  AUC(0-8h) Cycle 1 Day 1 | 2680 (894) | 2502 (994) | 1013 (733) |
  AUC(0-4h) Cycle 2 Day 1: number analyzed (Participants) | 4 | 2 | 3 | 28
  AUC(0-4h) Cycle 2 Day 1 | 3067 (1628) | 5615 (696) | 7375 (3818) | 1994 (797)

12. Secondary Outcome: Part 1 & 2: Measure Plasma Concentrations of Talazoparib.
Description: Plasma concentrations of talazoparib will be measured.
Time Frame: Part 1: Cycle 1 Day 15: Pre-dose; Parts 1& 2 Cycle 2 Day 1: Pre-dose; Cycle 2 Day 15: Pre-dose (each cycle is 28 days)
Population: Part 1 (All evaluable participants): C1D15; Parts 1 & 2 (All evaluable participants): C2D1 & C2D15
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 2 - Stages 1 and 2
Number analyzed (Participants) | 6 | 5 | 3 | 35
pg/mL
  Cycle 1 Day 15 Pre-dose: number analyzed (Participants) | 6 | 5 | 3 | 0
  Cycle 1 Day 15 Pre-dose | 4813.3 (2278.1) | 4582 (1562.5) | 5650 (2714.1) |
  Cycle 2 Day 1 Pre-dose: number analyzed (Participants) | 5 | 4 | 3 | 35
  Cycle 2 Day 1 Pre-dose | 3814 (3092) | 3584.3 (2819.4) | 8220 (4073.1) | 3129.8 (2190.2)
  Cycle 2 Day 15 Pre-dose: number analyzed (Participants) | 4 | 4 | 2 | 30
  Cycle 2 Day 15 Pre-dose | 3952.5 (1348.7) | 4892.5 (1957.5) | 4840 (3097.1) | 4240 (2110.4)

13. Secondary Outcome: Expansion Cohorts A, B, and C: Measure Plasma Concentrations of ZEN003694 and the Active Metabolite ZEN003791.
Description: Plasma concentrations of ZEN003694 and the active metabolite ZEN003791 will be measured.
Time Frame: Cycle 2 Day 1: Pre-dose, 1 hour, 2 hours, and 4 hours post-dose; Cycle 2 Day 15: Pre-dose (each cycle is 28 days)
Population: Cohorts A and B - Study was terminated prior to PK analysis for samples collected from cohorts A and B, therefore data was not obtained. Data will never be obtained and reported for this measure. Cohort C - All Evaluable Participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients | Expansion Cohort B - ZEN003694 Monotherapy | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients
Number analyzed (Participants) | 0 | 0 | 15
ng/mL
  ZEN003694 Cycle 2 Day 1 - Predose |  |  | 33.82 (21.4)
  ZEN003694 Cycle 2 Day 1 - 1 hour: number analyzed (Participants) | 0 | 0 | 10
  ZEN003694 Cycle 2 Day 1 - 1 hour |  |  | 383.9 (259.1)
  ZEN003694 Cycle 2 Day 1 - 2 hours: number analyzed (Participants) | 0 | 0 | 10
  ZEN003694 Cycle 2 Day 1 - 2 hours |  |  | 397.2 (232.4)
  ZEN003694 Cycle 2 Day 1 - 4 hours: number analyzed (Participants) | 0 | 0 | 10
  ZEN003694 Cycle 2 Day 1 - 4 hours |  |  | 345.3 (116.9)
  ZEN003694 Cycle 2 Day 15 - Predose: number analyzed (Participants) | 0 | 0 | 10
  ZEN003694 Cycle 2 Day 15 - Predose |  |  | 45.2 (28.6)
  ZEN003791 Cycle 2 Day 1 - Predose |  |  | 110.2 (84.3)
  ZEN003791 Cycle 2 Day 1 - 1 hour: number analyzed (Participants) | 0 | 0 | 10
  ZEN003791 Cycle 2 Day 1 - 1 hour |  |  | 231.0 (158.9)
  ZEN003791 Cycle 2 Day 1 - 2 hours: number analyzed (Participants) | 0 | 0 | 10
  ZEN003791 Cycle 2 Day 1 - 2 hours |  |  | 268.4 (207.0)
  ZEN003791 Cycle 2 Day 1 - 4 hours: number analyzed (Participants) | 0 | 0 | 10
  ZEN003791 Cycle 2 Day 1 - 4 hours |  |  | 303.8 (154.1)
  ZEN003791 Cycle 2 Day 15 - Predose: number analyzed (Participants) | 0 | 0 | 10
  ZEN003791 Cycle 2 Day 15 - Predose |  |  | 169.0 (111.3)

14. Secondary Outcome: Expansion Cohorts A and C: Measure Plasma Concentrations of Talazoparib.
Description: Plasma concentrations of talazoparib will be measured.
Time Frame: Cycle 2 Day 1: Pre-dose, Cycle 2 Day 15: Pre-dose (each cycle is 28 days)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients
Number analyzed (Participants) | 0 | 15
pg/mL
  Talazoparib Cycle 2 Day 1 - Pre-dose |  | 2152.8 (2031.9)
  Talazoparib Cycle 2 Day 15 - Pre-dose: number analyzed (Participants) | 0 | 10
  Talazoparib Cycle 2 Day 15 - Pre-dose |  | 4494.1 (3139.8)

15. Secondary Outcome: Part 2, Expansion Cohorts A and C: Change From Baseline in Global Health Status/Quality of Life (QoL) Measured by EORTC QLQ-C30 for Overall Duration
Description: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30): cancer-specific instrument with 30 questions to assess the participant QoL. First 28 questions used to evaluate 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, nausea and vomiting, pain) and other single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Each question assessed on 4-point scale (1= not at all, 2= a little, 3= quite a bit, 4= very much); functional scales: higher score = better level of functioning; symptom scale: higher score = more severe symptoms; for single items: higher score= more severe problem. Last 2 questions used to evaluate global health status (GHS)/QoL. Each question was assessed on 7-point scale (1= very poor to 7= excellent). Scores averaged, transformed to 0-100 scale; higher score=better quality of life/better level of functioning.
Time Frame: Screening and Day 1 of every 28-day Cycle, up to 18 months (Overall Duration)
Reporting Status: Not Posted

16. Secondary Outcome: Part 2, Expansion Cohorts A and C: Change From Baseline in Breast Symptoms Scale as Assessed by the EORTC-QLQ-BR23
Description: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Breast Cancer Module (EORTC-QLQ-BR23) is a disease-specific module for breast cancer developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer. EORTC-QLQ-BR23 symptoms subscale includes 4 items: systemic therapy side effects, breast symptoms, arm symptoms, upset by hair loss. Each item is rated by choosing 1 of 4 possible responses that record the level of intensity (1= not at all, 2= a little, 3= quite a bit, and 4= very much), higher scores=high level of symptom/problems.
Time Frame: Screening and Day 1 of every 28-day Cycle, up to 18 months (Overall Duration)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Cycle 1 Day 1 to 30 days post last dose (each cycle is 28 days) up to 22 months.
Description: Adverse events were collected in all participants. For an event to be recorded as an AE, the onset must occur during or after the patient's first exposure to study drug and no later than 30 days after the last study drug dose.
Groups:
- Expansion Cohort B - ZEN003694 Combination: Post cross-over to combination treatment of ZEN003694 48 mg PO QD with 0.75 mg Talazoparib PO QD at the time of disease progression (but no sooner than after 6 weeks of monotherapy). Patients have histologically confirmed Triple Negative Breast Cancer and have no documented germline mutations of BRCA1 or BRCA2. Includes sites in the US and EU.
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 2 Stages 1 & 2 | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients | Expansion Cohort B - ZEN003694 Monotherapy | Expansion Cohort B - ZEN003694 Combination | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/3 | 3/42 | 5/21 | 0/3 | 0/1 | 1/32
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/8 | 1/3 | 11/42 | 10/21 | 0/3 | 0/1 | 14/32
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 3/3 | 42/42 | 21/21 | 2/3 | 1/1 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Dose Escalation: Cohort 1 (N=6) | Part 1 Dose Escalation: Cohort 2 (N=8) | Part 1 Dose Escalation: Cohort 3 (N=3) | Part 2 Stages 1 & 2 (N=42) | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients (N=21) | Expansion Cohort B - ZEN003694 Monotherapy (N=3) | Expansion Cohort B - ZEN003694 Combination (N=1) | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients (N=32)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 7
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Dose Escalation: Cohort 1 (N=6) | Part 1 Dose Escalation: Cohort 2 (N=8) | Part 1 Dose Escalation: Cohort 3 (N=3) | Part 2 Stages 1 & 2 (N=42) | Expansion Cohort A - Combination Treatment in Post-TROP2-ADC Patients (N=21) | Expansion Cohort B - ZEN003694 Monotherapy (N=3) | Expansion Cohort B - ZEN003694 Combination (N=1) | Expansion Cohort C - Combination Treatment in TROP2-ADC-naïve Patients (N=32)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 8 | 10 | 0 | 0 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 8 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Dyschromatopsia (Eye disorders) | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 1
Photophobia (Eye disorders) | 1 | 1 | 0 | 3 | 2 | 0 | 0 | 1
Photopsia (Eye disorders) | 1 | 1 | 1 | 9 | 3 | 1 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 1 | 4 | 5 | 0 | 0 | 7
Visual impairment (Eye disorders) | 0 | 1 | 0 | 6 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 0 | 6 | 5 | 0 | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 6 | 2 | 1 | 0 | 5
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 3 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 5 | 0 | 19 | 11 | 0 | 0 | 19
Vomiting (Gastrointestinal disorders) | 2 | 4 | 0 | 11 | 4 | 1 | 0 | 13
Asthenia (General disorders) | 1 | 1 | 1 | 4 | 0 | 0 | 0 | 3
Fatigue (General disorders) | 4 | 3 | 1 | 14 | 13 | 0 | 0 | 7
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Pain (General disorders) | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 0 | 10 | 3 | 0 | 0 | 13
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 0 | 12 | 5 | 0 | 0 | 13
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 25
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 5 | 1 | 0 | 0 | 8
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 5
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 6
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 6 | 3 | 0 | 0 | 8
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | 4 | 2 | 0 | 1 | 12
Platelet count decreased (Investigations) | 3 | 4 | 0 | 16 | 8 | 1 | 1 | 16
Weight decreased (Investigations) | 2 | 1 | 1 | 2 | 1 | 0 | 0 | 6
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 12
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 1 | 11 | 7 | 0 | 0 | 18
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 6 | 8 | 0 | 0 | 19
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 3 | 0 | 0 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 5 | 0 | 0 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 5 | 5 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 3
Dysgeusia (Nervous system disorders) | 2 | 1 | 1 | 9 | 5 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 5 | 3 | 0 | 0 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 3 | 0 | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 5 | 3 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0 | 8 | 3 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure permission may only be granted upon sponsor review.

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT03901469/Prot_002.pdf
  • Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03901469/SAP_003.pdf